CLINICAL TRIAL: NCT05785169
Title: Ending the HIV Epidemic: An All-facility Intervention for Patient and Healthcare Staff Well-being
Brief Title: Ending the HIV Epidemic for Patient and Healthcare Staff Well-being
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Rutgers University (Other); Florida State University (Other); RTI International (Other); Duke University (Other)
Responsible Party: Principal Investigator, Corina Lelutiu-Weinberger, Associate Professor of Health Sciences Research, Columbia University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAU1559; 1R01NR020583 (NIH)
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Stigma; HIV; Well-Being, Psychological
MeSH Terms: conditions — Social Stigma; Psychological Well-Being | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The intervention will be implemented across three steps with a total of 6 clinics (2 clinics per step). This stepped-wedge design will use stratified randomization to assign the timing of the intervention to one of 3 study sequences. Clinics would have been selected based on high rates of HIV. The criterion used to randomize clinics (by strata) to one of the 3 study sequences will be urbanicity (rural/suburban vs urban), which accounts for clinic size (# patients/year). Within each of the 2 strata, 3 clinics will be randomized to one of the 3 groups of clusters. Stratified Randomization will be conducted in Statistical Analysis System (SAS).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- First Cluster (Experimental): The intervention will be implemented across three steps with a total of 6 clinics (two clinics per step). The earliest roll-out of the intervention will be at the clinics randomized to Cluster 1.
  The intervention consists of a mix of Workshops, Interactive Trainings and Learning Circles (virtual and in-person). In the first workshop, the investigators will present baseline findings to all clinic members to 1) raise awareness for the need for intervention to reduce stigma, 2) facilitate collaborative processes, 3) catalyze change for practice change, to 4) guide the intervention process. This workshop will be followed by a series of interactive trainings covering relevant topics, and the creation of a manual to guide the implementation and sustainability of stigma reduction efforts.
  Interventions: Behavioral: All-facility Training
- Second Cluster (Experimental): The intervention will be implemented across three steps with a total of 6 clinics (two clinics per step). The earliest roll-out of the intervention will be at the clinics randomized to Cluster 1.
  The intervention consists of a mix of Workshops, Interactive Trainings and Learning Circles (virtual and in-person). In the first workshop, the investigators will present baseline findings to all clinic members to 1) raise awareness for the need for intervention to reduce stigma, 2) facilitate collaborative processes, 3) catalyze change for practice change, to 4) guide the intervention process. This workshop will be followed by a series of interactive trainings covering relevant topics, and the creation of a manual to guide the implementation and sustainability of stigma reduction efforts.
  Interventions: Behavioral: All-facility Training
- Third Cluster (Experimental): The intervention will be implemented across three steps with a total of 6 clinics (two clinics per step). The earliest roll-out of the intervention will be at the clinics randomized to Cluster 1.
  The intervention consists of a mix of Workshops, Interactive Trainings and Learning Circles (virtual and in-person). In the first workshop, the investigators will present baseline findings to all clinic members to 1) raise awareness for the need for intervention to reduce stigma, 2) facilitate collaborative processes, 3) catalyze change for practice change, to 4) guide the intervention process. This workshop will be followed by a series of interactive trainings covering relevant topics, and the creation of a manual to guide the implementation and sustainability of stigma reduction efforts.
  Interventions: Behavioral: All-facility Training

INTERVENTIONS:
Behavioral: All-facility Training — The HP+ curriculum includes total-site training and co-facilitation via participatory modules. To change clinic culture, a multi-level approach that includes the whole facility and reaches all parties is required. The intervention aims to modify top-down mechanisms of influence. The training is modeled on these principles and supports the development of multiple stigma-reduction strategies to improve patient and staff wellbeing.
  Other Names: Health Policy+ infused with US HIV care clinic-relevant content and activities

SUMMARY:
The scope of this study is to engage Ryan White HIV/AIDS Program (RWHAP) funded organizations in the South/East US to co-develop context-responsive programs utilizing evidence-informed interventions to reduce stigma against living with HIV (PLH) who have difficulties accessing and remaining engaged in life-saving treatment. Six RWHAP clinics will be selected to participate and be assigned to one of three sequences (two clinics per cluster). All members will complete participate in interactive trainings to raise awareness of and reduce stigma, from the clinic policy level to individual attitudes. All clinic members and select patients will complete self-administered surveys every 6 months over 24 months.

DETAILED DESCRIPTION:
The scope of this study is to engage Ryan White HIV/AIDS Program (RWHAP) funded organizations in the South/East US to co-develop context-responsive programs utilizing evidence-informed interventions to reduce stigma against living with HIV (PLH) who have difficulties accessing and remaining engaged in life-saving treatment. The proposed intervention draws on the evidence-based Health Policy Plus (HP+) 'total' facility HIV stigma-reduction intervention and Contact Theory, which have demonstrated efficacy in improving inter-group relations. The program targets the clinics' organizational and systems levels to affect patient outcomes and staff wellbeing, at the individual level. In Aim 1, we will rigorously select 6 clinics in the South/East US. In Aim 2, after a baseline assessment (N=180), we will conduct a stepped wedge cluster randomized trial of the stigma reduction intervention. At each of the 3 steps, two randomized clinics will receive the training, which will support clinics to 1) identify/create organizational-level anti-stigma policies and practices to reduce stigma, and 2) deliver participatory trainings to all staff. Each cluster will receive the intervention for 6 months, starting with Cluster Group 1, followed by Cluster Groups 2 and 3. In Aim 3, we will evaluate multi-level outcomes using the Consolidated Framework for Implementation Research (CFIR), including within the organization (primary outcome of Stigma Reduction Index - ratings of mission/vision statements, policies], clinic environment), systems (secondary outcomes of provider/staff attitudes; behavior), and individual patient level (tertiary outcomes of clinic-level HIV indicators, reports of stigmatization, clinic climate, anxiety, depression) outcomes. Assessments will take place every 6 months, with the clinics randomized to the second or third step having multiple assessments before the intervention. Patients at the clinics will be surveyed at each assessment (N=2,100). Findings will yield a manual for implementing total-facility stigma-reduction processes and content. Other RWHAP-funded clinics and facilities may be able to adopt this manualized, yet highly adaptable intervention packet.

ELIGIBILITY:
Inclusion Criteria:

* Selected Ryan White Clinics. Selection based on the following:

First, clinic leaders will complete a 15-min Site Characteristics Survey, assessing suitability for participation and clinic comparability for randomization purposes. Staff and leadership at Ryan White clinics will next complete an anonymous 15-minute Eligibility Survey.

Within each clinic, both clinic staff and patients will be invited to participate.

Exclusion Criteria:

* Non-Ryan White Clinics
* Clinics not located in the geographical area of interest
* Clinics that are not interested in participating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change in Stigma Index (SI) | Baseline, 6, 12, 18, and 24 months
  The SI is a rating of clinic mission/vision statements, the anti-stigma policy, and the clinic context. A change in the mean score of SI post-intervention implementation will be measured. Scores range from 0-100, with a higher score indicating increased anti-stigma policies and procedures.

SECONDARY OUTCOMES:
Change in Cultural Humility Score | Baseline, 6, 12, 18, and 24 months
  Cultural humility as measured by the adapted Trauma-Informed, Resilience-Oriented Care (TI-ROC) Cultural Humility Scale, which assess staff's perceptions of colleagues and clinic context. Scores range from 12-60. The negative items are reverse coded such that higher scores indicate higher cultural humility indicating better outcomes.

OTHER OUTCOMES:
Change in Time to Linkage to Care | Baseline, 6, 12, 18, and 24 months
  Change in time to linkage to care from diagnosis at the clinics.
Change in Patients Retained in Care | Baseline, 6, 12, 18, and 24 months
  Change in the number of patients retained in care at the clinics.
Change in Number of Patients HIV Virally Suppressed | Baseline, 6, 12, 18, and 24 months
  Change in the number of patients virally suppressed at the clinics. Viral suppression defined as less than 200 copies/mL.
Change in Frequency of Perceived HIV and Other Stigmas | Baseline, 6, 12, 18, and 24 months
  Change in the frequency of perceived stigma-related events by staff and patients attending the clinic as collected by self-administered Experiences of Perceived Stigma survey.
Change in Depression and Anxiety | Baseline, 6, 12, 18, and 24 months
  A 4-item scale that assesses depression and anxiety (PHQ-4) over the past week. Scores range from 0-63 with a lower score indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Corina Lelutiu-Weinberger, PhD, Principal Investigator — Columbia University; Felicia A Browne, ScD, Principal Investigator — RTI International
Locations (1):
- Columbia University School of Nursing, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No